CLINICAL TRIAL: NCT01048333
Title: A Randomised, Placebo-controlled, Double-blind (Double-dummy Technique),Crossover, Multi-centre Study, to Evaluate Onset of Effect in Patients With Chronic Obstructive Pulmonary Disease (COPD) Treated With Formoterol Turbuhaler® 9 μg, Compared With Serevent® Diskus® 50 μg.
Brief Title: Evaluate Onset of Effect in Patients With Chronic Obstructive Pulmonary Disease (COPD) Treated With Formoterol Turbuhaler®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5127C00001
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Onset of effect; COPD; Oxis Turbuhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Formoterol, then Salmeterol, then Placebo (Experimental): Formoterol Turbuhaler 9 μg and Placebo Diskus first, then Salmeterol Diskus 50 μg and Placebo Turbuhaler, then Placebo Diskus and Placebo Turbuhaler
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo
- Salmeterol, then Palcebo, then Formoterol (Experimental): Salmeterol Diskus 50 μg and Placebo Turbuhaler first, then Placebo Diskus and Placebo Turbuhaler, then Formoterol Turbuhaler 9 μg and Placebo Diskus
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo
- Placebo, then Formoterol, then Salmeterol (Experimental): Placebo Diskus and Placebo Turbuhaler first,then Formoterol Turbuhaler 9 μg and Placebo Diskus, then Salmeterol Diskus 50 μg and Placebo Turbuhaler
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo
- Formoterol, then Placebo, then Salmeterol (Experimental): Formoterol Turbuhaler 9 μg and Placebo Diskus first, then Placebo Diskus and Placebo Turbuhaler, then Salmeterol Diskus 50 μg and Placebo Turbuhaler
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo
- Salmeterol, then Formoterol, then Placebo (Experimental): Salmeterol Diskus 50 μg and Placebo Turbuhaler first, then Formoterol Turbuhaler 9 μg and Placebo Diskus, then Placebo Diskus and Placebo Turbuhaler
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo
- Placebo, then Salmeterol, then Formoterol (Experimental): Placebo Diskus and Placebo Turbuhaler first, then Salmeterol Diskus 50 μg and Placebo Turbuhaler, then Formoterol Turbuhaler 9 μg and Placebo Diskus
  Interventions: Drug: Formoterol; Drug: Salmeterol; Drug: Placebo

INTERVENTIONS:
Drug: Formoterol — Formoterol Turbuhaler 9 μg and Placebo Diskus
Drug: Salmeterol — Salmeterol Diskus 50 μg and Placebo Turbuhaler
Drug: Placebo — Placebo Diskus and Placebo Turbuhaler

SUMMARY:
* Primary objective is to evaluate time to onset of effect of formoterol, 9 μg single dose,compared with salmeterol, 50 μg single dose, in patients with moderate COPD.Forced Expiratory Volume in 1 second (FEV1) measured by spirometry 5 minutes postdose.
* Secondary efficacy variables: Average FEV1 during the first 15 minutes (area under the FEV1 curve from 0 to 15 minutes), Average FEV1 during 120 minutes (area under the FEV1 curve from 0 to 120 minutes)

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD according to GOLD guidelines, and current COPD symptoms
* A current or previous smoking history equivalent to 10 or more packs per year (1 pack year = 20 cigarettes smoked per day for one year).
* Documented use of a short-acting inhaled bronchodilator (β2-agonist or anticholinergics) as reliever medication.

Exclusion Criteria:

* A history and/or current diagnosis of asthma.
* Patients who have experienced COPD exacerbation requiring hospitalisation and/or a course of antibiotics and/or a course of systemic steroid within 30 days (from end of exacerbation treatment) prior to Visit 1 and/or during the run-in period.
* A history and/or current diagnosis of atopic diseases such as allergic rhinitis or eczema before the age of 40.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Cazzola, professor, Principal Investigator — Italy; Georgios Stratelis, Study Director — AstraZeneca MC Sweden
Locations (17):
- Italy (10):
  - Research Site, Bussolengo
  - Research Site, Cassano delle Murge
  - Research Site, Catanzaro
  - Research Site, Cava de' Tirreni
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Prato
  - Research Site, Roma
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Lund

REFERENCES:
- [Derived] Cazzola M, Paggiaro P, Palange P, Bjermer L, Ausin P, Carlsson LG, Ekelund J, Lotvall J. Onset of action of formoterol versus salmeterol via dry powder inhalers in moderate chronic obstructive pulmonary disease: a randomized, placebo-controlled, double-blind, crossover study. Clin Drug Investig. 2012 Mar 1;32(3):147-55. doi: 10.2165/11630880-000000000-00000. PMID 22235841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at 14 clinics in 3 countries: Sweden (4 clinics); Italy (6 clinics); Spain (6 clinics)between January and May 2010
Pre-assignment Details: 141 patients enrolled; 32 excluded: 28 due to eligibility criteria not fulfilled and 4 for subject decision
Period: Treatment Period 1
Arm/Group | Formoterol, Then Salmeterol, Then Placebo | Salmeterol, Then Palcebo, Then Formoterol | Placebo, Then Formoterol, Then Salmeterol | Formoterol, Then Placebo, Then Salmeterol | Salmeterol, Then Formoterol, Then Placebo | Placebo, Then Salmeterol, Then Formoterol
Started | 21 | 19 | 16 | 18 | 17 | 18
Completed | 21 | 19 | 16 | 18 | 17 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-Out Period 1 of 2 - 7 Days
Arm/Group | Formoterol, Then Salmeterol, Then Placebo | Salmeterol, Then Palcebo, Then Formoterol | Placebo, Then Formoterol, Then Salmeterol | Formoterol, Then Placebo, Then Salmeterol | Salmeterol, Then Formoterol, Then Placebo | Placebo, Then Salmeterol, Then Formoterol
Started | 21 | 19 | 16 | 18 | 17 | 18
Completed | 21 | 19 | 16 | 18 | 17 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Formoterol, Then Salmeterol, Then Placebo | Salmeterol, Then Palcebo, Then Formoterol | Placebo, Then Formoterol, Then Salmeterol | Formoterol, Then Placebo, Then Salmeterol | Salmeterol, Then Formoterol, Then Placebo | Placebo, Then Salmeterol, Then Formoterol
Started | 21 | 19 | 16 | 18 | 17 | 18
Completed | 21 | 19 | 16 | 18 | 17 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-Out Period 2 of 2 - 7 Days
Arm/Group | Formoterol, Then Salmeterol, Then Placebo | Salmeterol, Then Palcebo, Then Formoterol | Placebo, Then Formoterol, Then Salmeterol | Formoterol, Then Placebo, Then Salmeterol | Salmeterol, Then Formoterol, Then Placebo | Placebo, Then Salmeterol, Then Formoterol
Started | 21 | 19 | 16 | 18 | 17 | 18
Completed | 21 | 18 | 16 | 18 | 17 | 18
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Formoterol, Then Salmeterol, Then Placebo | Salmeterol, Then Palcebo, Then Formoterol | Placebo, Then Formoterol, Then Salmeterol | Formoterol, Then Placebo, Then Salmeterol | Salmeterol, Then Formoterol, Then Placebo | Placebo, Then Salmeterol, Then Formoterol
Started | 21 | 18 | 16 | 18 | 17 | 18
Completed | 21 | 18 | 16 | 18 | 17 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all 3 arms : Formoterol, Salmeterol and Placebo.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 109
Age Continuous [Mean (Full Range); unit: years] | 66.5 [41.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 81

OUTCOME MEASURES:

1. Primary Outcome: FEV1(Forced Expiratory Volume in 1 Second) Measured by Spirometry 5 Minutes Post Dose
Description: FEV1(Forced Expiratory Volume in 1 second) measured by spirometry 5 minutes post dose, percentage change versus pre dose FEV1
Time Frame: Pre-dose and 5 minutes post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Groups:
- Formoterol: Formoterol Turbuhaler 9 mcg
- Salmeterol: Serevent Diskus (salmeterol) 50 mcg
- Placebo: Placebo salmeterol Diskus and Placebo Turbuhaler
Arm/Group | Formoterol | Salmeterol | Placebo
Number analyzed (Participants) | 108 | 109 | 109
percentage change | 1.072 [1.055 to 1.088] | 1.041 [1.025 to 1.057] | 1.007 [0.992 to 1.023]

2. Secondary Outcome: Average FEV1 During the First 15 Minutes Post Dose
Description: Average FEV1 during the first 15 minutes post dose, change versus pre dose FEV1
Time Frame: Pre dose and 15 minutes post dose
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Formoterol | Salmeterol | Placebo
Number analyzed (Participants) | 108 | 109 | 109
percentage change | 1.064 [1.052 to 1.077] | 1.041 [1.030 to 1.053] | 1.012 [1.001 to 1.024]

3. Secondary Outcome: Average FEV1 During 120 Minutes Post Dose
Description: Average FEV1 during 120 minutes post dose, change versus pre dose FEV1
Time Frame: Pre dose and 120 minutes post dose
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Formoterol | Salmeterol | Placebo
Number analyzed (Participants) | 108 | 109 | 109
percentage change | 1.096 [1.079 to 1.112] | 1.082 [1.066 to 1.098] | 1.014 [0.999 to 1.029]

4. Secondary Outcome: Percentage of Patients Who Has Achieved at Least 12 % Increase in FEV1
Description: Percentage of patients who has achieved at least 12 % increase in FEV1 at each time point between 5 to 120 minutes post dose, change versus pre dose FEV1
Time Frame: Pre dose, 5, 10, 15, 20, 30, 40, 50, 60 and 120 minutes post dose
Measure: Number; unit: Percentage of Participants
Arm/Group | Formoterol | Salmeterol | Placebo
Number analyzed (Participants) | 108 | 109 | 109
Percentage of Participants
  5 min | 23.1 | 9.2 | 6.4
  10 min | 38.0 | 17.6 | 7.3
  15 min | 39.8 | 23.9 | 9.2
  20 min | 44.4 | 27.5 | 10.1
  30 min | 45.4 | 32.1 | 13.8
  40 min | 49.1 | 36.7 | 15.6
  50 min | 53.7 | 40.4 | 16.5
  60 min | 54.6 | 43.1 | 18.3
  120 min | 55.6 | 48.6 | 20.2
Statistical Analysis 1: Comparison: Formoterol vs Salmeterol; Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 2.090, 95% CI 2-sided [1.31 to 3.35]
Statistical Analysis 2: Comparison: Formoterol vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 6.534, 95% CI 2-sided [3.55 to 12.02]
Statistical Analysis 3: Comparison: Salmeterol vs Placebo; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 3.127, 95% CI 2-sided [1.77 to 5.52]

5. Secondary Outcome: Adverse Events
Description: Number of participants with at least 1 AE.
Time Frame: At baseline and at each day of treatment
Measure: Number; unit: Participants
Arm/Group | Formoterol | Salmeterol | Placebo
Number analyzed (Participants) | 108 | 109 | 109
Participants | 6 | 6 | 2

ADVERSE EVENTS:
Arm/Group | Formoterol | Salmeterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/109 | 0/109
Other Adverse Events (participants affected / at risk) | 0/108 | 0/109 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less